CLINICAL TRIAL: NCT01582776
Title: A Phase Ib/II Study of OBINUTUZUMAB Combined to LENALIDOMIDE for the Treatment of Follicular and Relapsed/Refractory Aggressive (DLBCL and MCL) B-cell Lymphoma
Brief Title: Study of OBINUTUZUMAB Combined to LENALIDOMIDE for the Treatment of Relapsed/Refractory Follicular and Aggressive B-cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GALEN
Record Dates: First submitted 2012-04-20; First posted 2012-04-23 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Follicular Lymphoma Patients (Phase IB); Follicular and Agressive (DLBCL&MCL) B-cell Lymphoma Patients (Phase II)
MeSH Terms: interventions — Lenalidomide; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide and GA101 (Experimental): Ga101 and lenalidomide
  Interventions: Drug: Lenalidomide and GA101

INTERVENTIONS:
Drug: Lenalidomide and GA101 — 1000mg of GA101 on D8, D15 and D22of cycle 1 and on D1 of cycles 2 to 6. Oral lenalidomide once daily at 10/15/20/25mg (phase I part) or at recommended dose (phase II part) on days 1 to 21 of a 28-day cycle for the first cycle and on days 2 to 22 of a 28-day cycle for cycles 2 to 6.
  Other Names: Revlimid; Obinutuzumab

SUMMARY:
This study is to determine first the appropriate dose of lenalidomide to administer in combination with fixed doses of obinutuzumab in relapsed/refractory follicular lymphoma patients.

In a second step, this study aims to determine the efficacy of this combination in 3 separate populations: relapsed/refractory aggressive lymphoma (diffuse large B-cell lymphoma and mantle cell lymphoma: cohort 1), relapsed/refractory follicular lymphoma (cohort 2) and previously untreated follicular lymphoma (cohorts 3 and 4).

DETAILED DESCRIPTION:
This study is an open label, multicenter study with two phases:

The Phase IB part of the study is a dose escalation study of lenalidomide (Revlimid) administered orally during on 3 weeks of every 28-day cycle, in combination with fixed doses of obinutuzumab (GA101) in relapsed/refractory follicular lymphoma patients.

The Phase II part of the study is an efficacy study of the association of the recommended dose of lenalidomide associated with GA101 in 2 separate populations of patients: relapsed/refractory aggressive lymphoma (diffuse large B-cell lymphoma and mantle cell lymphoma: cohort 1), relapsed/refractory follicular lymphoma (cohort 2) and previously untreated follicular lymphoma (cohorts 3 and 4). First, all patients will receive a combination of obinutuzumab and lenalidomide for a total of 6 cycles. Patients who achieve at least a partial response after 6 cycles will receive a maintenance treatment with obinutuzumab for 2 years and Lenalidomide for 1 year as tolerated, or until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Phase IB only: Histologically documented CD20-positive follicular lymphoma (WHO grade 1, 2, or 3a) patients
* Phase II: Patients with either histologically documented CD20-positive Diffuse large-cell lymphoma or Mantle cell lymphoma (cohort 1) or follicular lymphoma, WHO grade 1, 2 or 3a (cohort 2-3-4)
* Phase IB and II:
* Relapsed/refractory NHL after ≥1 prior R-containing regimen with no curative option (cohort 2 only)
* Aged 18 years or more
* ECOG performance status 0, 1 or 2
* At least one bi-dimensionally measurable nodal or tumor lesion defined by CT scan as: greatest transverse diameter > 1.5 cm and a short axis ≥ 10mm
* Signed inform consent
* Life expectancy ≥ 3 months.
* All subjects must be able to understand and fulfill the lenalidomide Pregnancy Prevention Plan requirements (see in appendix)
* Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual contact during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; 3) dose interruptions; and 4) for at least 2 months after discontinuation of all study treatments.

Exclusion Criteria:

* Previous treatment with obinutuzumab or lenalidomide
* Known CD20 negative status at relapse/progression. Biopsy at relapse/progression is recommended but not mandatory
* Central nervous system or meningeal involvement by lymphoma
* Contraindication to any drug contained in the study treatment regimen
* Known HIV or HTLV-1 infection, positive serology to HB surface antigen [HBsAg] or total HB core antibody [anti-HB-c]) and Hepatitis C (Hepatitis C virus [HCV] antibody)
* Any serious active disease or co-morbid medical condition (such as New York Heart Association Class II or IV cardiac disease, severe arrhythmia, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina) or pulmonary disease (including obstructive pulmonary disease and history of bronchospasm or other according to investigator's decision)
* Any of the following laboratory abnormalities unless secondary to underlying lymphoma:

  * Absolute neutrophil count (ANC) < 1,500 cells/mm3 (1.5 x 109/L).
  * Platelet count < 100,000/mm3 (100 x 109/L) unless due to lymphoma for phase II part.
  * Serum SGOT/AST or SGPT/ALT 3.0 x upper limit of normal (ULN) unless disease involvement.
  * Serum total bilirubin > 2.0 mg/dL (34 μmol/L), except if disease related or in case of Gilbert syndrome
  * Calculated creatinine clearance (Cockcroft-Gault formula or MDRD) of < 50 mL /min. For phase II part of the study, patients with calculated creatinine clearance between 30 and 50ml/min can be included and lenalidomide dose will be adjusted as follows (10mg once daily)
* Prior history of malignancies other than lymphoma unless the subject has been free of the disease for ≥ 5 years
* Any serious medical condition, laboratory abnormality (other than mentioned above), or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or lactating females.
* Prior ≥ Grade 3 allergic reaction/hypersensitivity to thalidomide.
* Prior ≥ Grade 3 rash or any desquamating (blistering) rash while taking thalidomide.
* Subjects with ≥ Grade 2 neuropathy.
* Use of any standard or experimental anti-cancer drug therapy within 28 days of the initiation (Day 1) of study drug therapy
* Patients taking corticosteroids during 4 weeks before inclusion, unless administered at a dose equivalent to ≤ 10 mg/day prednisone (over these 4 weeks)
* Prior history of Progressive Multifocal Leukoencephalopathy (PML)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2012-10-03 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Phase I part: Determination of the recommended dose of lenalidomide in combination with fixed doses of GA101 | 28 days
  The determination of the recommended dose of lenalidomide in combination with fixed doses of GA101 will be performed by a dose escalation approach. Dose Limiting Toxicities (DLTs) observed during the administration of the first 2 cycles of the study will be listed for each escalation step.
Phase II part: Overall Response Rate (CR+CRu+PR) after 6 cycles | 24 weeks
  Response rates at the end of treatment including maintenance will be expressed as percentages with their 95% Exact Clopper Pearson Confidence Interval limits

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 4.5 years
  Overall survival will be measured from the date of inclusion to the date of death from any cause.
  Alive patients will be censored at their last date known to be alive
Event Free survival | Up to 4.5 years
  Event-Free Survival will be measured from the date of inclusion to the date of first documented disease progression, relapse, initiation of new anti-lymphoma therapy or death from any cause.
Progression free survival | Up to 4.5 years
  Progression-Free Survival will be measured according to the Cheson 2007 criteria. Responding patients and patients who are lost to follow up will be censored at their last tumor assessment date.
Response duration | Up to 4.5 years
  Patients alive and free of progression will be censored at their last follow-up date
Response rate at the end of maintenance treatment | 2.5 years
  Response rates will be evaluated at the end of maintenance phase for patients who achieve a CR/PR after induction treatment and received at least one dose of maintenance. Assessment of response will be based on the International Workshop to Standardize Response criteria for NHL (Criteria for evaluation of response in Non-Hodgkin's lymphoma (Cheson, 2007)). Patient without response assessment after maintenance treatment (due to whatever reason) will be considered as non-responder.
Complete response rate after induction | 24 weeks
  Disease response evaluation after 6 cycles will be used to determine the Complete Response Rate. Response after 6 cycles will be assessed only if patient completes induction phase. Assessment of response will be based on the International Workshop to Standardize Response criteria for NHL (Criteria for evaluation of response in Non-Hodgkin's lymphoma (Cheson, 1999 and 2007)).
Complete response rate after 3 cycles | 12 weeks
  Disease response evaluation after 3 cycles will be used to determine the Complete Response Rate.
  Response after 3 cycles will be assessed at the end of completion of the 3 cycles if patient received all 3 cycles or at withdrawal. Assessment of response will be based on the International Workshop to Standardize Response criteria for NHL (Criteria for evaluation of response in Non-Hodgkin's lymphoma (Cheson, 1999 and 2007).

CONTACTS AND LOCATIONS:
Overall Officials: Franck MORSCHHAUSER, Professor, Principal Investigator — Lymphoma Study Association; Roch HOUOT, Professor, Principal Investigator — Lymphoma Study Association
Locations (25):
- Belgium (7):
  - ZNA Stuivenberg, Antwerp
  - A.Z. Sint Jan AV, Bruges
  - institut Jules Bordet, Brussels
  - Université Catholique de Louvain Saint Luc, Brussels
  - AZ Groeninge - Campus Maria's Voorzienigheid, Kortrijk
  - CHU de Liège, Liège
  - Université Catholique de Louvain Mont Godinne, Yvoir
- France (18):
  - CHU d'Amiens, Amiens
  - Institut Bergonié, Bordeaux
  - Institut d'Hématologie de Basse Normandie, Caen
  - CHU d'Estaing, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHRU de Lille, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmette, Marseille
  - CHU St Eloi, Montpellier
  - CHU Brabois, Nancy
  - CHU Hôtel Dieu, Nantes
  - Hôpital St Louis, Paris
  - Centre François Magendie, Pessac
  - CH Lyon Sud, Pierre-Bénite
  - CHU Pontchaillou, Rennes
  - Centre henri Becquerel, Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bachy E, Houot R, Feugier P, Bouabdallah K, Bouabdallah R, Virelizier EN, Maerevoet M, Fruchart C, Snauwaert S, Le Gouill S, Marolleau JP, Molina L, Molucon-Chabrot C, Thieblemont C, Tilly H, Bijou F, Haioun C, Van den Neste E, Fabiani B, Meignan M, Cartron G, Salles G, Casasnovas O, Morschhauser F. Obinutuzumab plus lenalidomide in advanced, previously untreated follicular lymphoma in need of systemic therapy: a LYSA study. Blood. 2022 Apr 14;139(15):2338-2346. doi: 10.1182/blood.2021013526. PMID 34936697
- [Derived] Morschhauser F, Le Gouill S, Feugier P, Bailly S, Nicolas-Virelizier E, Bijou F, Salles GA, Tilly H, Fruchart C, Van Eygen K, Snauwaert S, Bonnet C, Haioun C, Thieblemont C, Bouabdallah R, Wu KL, Canioni D, Meignin V, Cartron G, Houot R. Obinutuzumab combined with lenalidomide for relapsed or refractory follicular B-cell lymphoma (GALEN): a multicentre, single-arm, phase 2 study. Lancet Haematol. 2019 Aug;6(8):e429-e437. doi: 10.1016/S2352-3026(19)30089-4. Epub 2019 Jul 8. PMID 31296423
- [Derived] Morschhauser F, Salles G, Le Gouill S, Tilly H, Thieblemont C, Bouabdallah K, Fabiani B, Menard C, Tarte K, Cartron G, Houot R. An open-label phase 1b study of obinutuzumab plus lenalidomide in relapsed/refractory follicular B-cell lymphoma. Blood. 2018 Oct 4;132(14):1486-1494. doi: 10.1182/blood-2018-05-853499. Epub 2018 Aug 1. PMID 30068505
- See also: Lymphoma Study Association — http://www.lysa-lymphoma.org/